CLINICAL TRIAL: NCT01845207
Title: Frailty Assessment Before Cardiac Surgery & Transcatheter Interventions
Status: Completed | Type: Observational
Sponsor: Jewish General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Duke University (Other); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other); Massachusetts General Hospital (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); McMaster University (Other); Montreal Heart Institute (Other); Royal Victoria Hospital, Canada (Other); St. Boniface Hospital (Other); Unity Health Toronto (Other); St. Paul's Hospital, Canada (Other); Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Jonathan Afilalo, MD MSc FACC FRCPC, Jewish General Hospital
Other Study IDs: MOP-123314
Record Dates: First submitted 2013-04-26; First posted 2013-05-03 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Aortic Stenosis; Cardiac Valve Replacement Complication; Fragility
Keywords: Aortic stenosis; Aortic valve replacement; Transcatheter aortic valve implantation; Outcomes; Frailty; Elderly
MeSH Terms: conditions — Aortic Valve Stenosis; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Tissue specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aortic valve replacement: Patients aged ≥70 years referred for surgical or transcatheter aortic valve replacement.

SUMMARY:
Frailty is a state of decreased physiologic reserves and vulnerability to stressors. Several tools exist to measure frailty, some based on physical tests and others on questionnaires, yet there is no agreement on which tool to recommend. This multi-center prospective cohort study is aimed at comparing various frailty assessment tools to determine which best predicts death or major complications after cardiac surgery or transcatheter intervention. The population of interest is elderly patients with severe aortic stenosis undergoing surgical or transcatheter aortic valve replacement. The frailty assessment tools under investigation include composite frailty scales, physical performance tests, muscle mass, and biomarker expression. The overall objective is to improve our ability to predict risk by measuring frailty using the optimal tool in elderly cardiovascular patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥70 years (a site-specific substudy at the JGH will enroll ages ≥21 years)
2. Severe AS
3. Referred for surgical or transcatheter AVR (with or without concomitant revascularization)
4. Signed informed consent

Exclusion Criteria:

1. Emergency surgery
2. Clinical instability: decompensated heart failure, active ischemia, unstable vital signs
3. Severe neuropsychiatric impairment
4. Not English or French speaking
5. Replacement of >1 valve or aortic surgery

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: In-patients and out-patients referred for surgical or transcatheter aortic valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Post-procedural mortality or major morbidity | 30 days
  Mortality is defined as death from any cause. Major morbidity is defined as an aggregate of the Society of Thoracic Surgeons (STS) and Valve Academic Research Consortium (VARC) composite endpoints. Additionally, the individual components of this composite endpoint will be examined.

SECONDARY OUTCOMES:
All-cause mortality | 6-12 months
Functional status | 6-12 months
Length of stay | 30 days

OTHER OUTCOMES:
Cognitive function | 6-12 months
Mood disturbance | 6-12 months
Delirium | 30 days
Disposition | 30 days
Readmission | 6-12 months
Cost analysis and resource use | 30 days
Echocardiographic function of ventricles and valves | 30 days
Longitudinal recovery of physical and cognitive functioning | Monthly (1-12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Afilalo, MD MSc, Principal Investigator — Jewish General Hospital
Locations (14):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
- Canada (9):
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Hamilton General Hospital, Hamilton, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Centre Hospitalier Universite de Montreal, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
- Hôpital Jacques Cartier, Massy, France

REFERENCES:
- [Derived] Shi SM, Sung M, Afilalo J, Lipsitz LA, Kim CA, Popma JJ, Khabbaz KR, Laham RJ, Guibone K, Lee J, Marcantonio ER, Kim DH. Delirium Incidence and Functional Outcomes After Transcatheter and Surgical Aortic Valve Replacement. J Am Geriatr Soc. 2019 Jul;67(7):1393-1401. doi: 10.1111/jgs.15867. Epub 2019 Mar 18. PMID 30882905
- [Derived] Afilalo J, Lauck S, Kim DH, Lefevre T, Piazza N, Lachapelle K, Martucci G, Lamy A, Labinaz M, Peterson MD, Arora RC, Noiseux N, Rassi A, Palacios IF, Genereux P, Lindman BR, Asgar AW, Kim CA, Trnkus A, Morais JA, Langlois Y, Rudski LG, Morin JF, Popma JJ, Webb JG, Perrault LP. Frailty in Older Adults Undergoing Aortic Valve Replacement: The FRAILTY-AVR Study. J Am Coll Cardiol. 2017 Aug 8;70(6):689-700. doi: 10.1016/j.jacc.2017.06.024. Epub 2017 Jul 7. PMID 28693934